CLINICAL TRIAL: NCT05626569
Title: Phase 2 Study of Anti-PD-1 Immunotherapy Combined With Stereotactic Body Radiation Therapy for Patients With Oligometastatic Esophageal Squamous Cell Carcinoma
Brief Title: Anti-PD-1 Immunotherapy Combined With SBRT for Patients With Oligometastatic ESCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Mian XI, MD, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-FXY-119
Record Dates: First submitted 2022-11-17; First posted 2022-11-23 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Esophageal Squamous Cell Carcinoma; Oligometastatic Disease
Keywords: esophageal cancer; oligometastases; PD-1; SBRT
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Esophageal Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PD-1 combined with SBRT for metastatic lesions (Experimental): Participants will receive anti-PD1 and SBRT to the metastatic lesions which are amenable to the delivery of SBRT after 4~6 cycles of systemic chemotherapy and anti-PD-1. SBRT for the metastatic lesions shall be conducted within two months after the completion of systemic therapy. The prescription of SBRT is determined by the investigator and the BED is required to over 50Gy.
  Interventions: Drug: PD-1 combined with SBRT

INTERVENTIONS:
Drug: PD-1 combined with SBRT — Anti-PD1 monoclonal antibody combined with SBRT. The SBRT defined as the radiation prescription with single dose equal or over 4Gy and the fractions less or equal to 10 fractions. BED equal or over 50Gy is required.
  Other Names: SBRT

SUMMARY:
The goal of this phase II clinical trial is to explore the efficacy and safety of anti-PD1 combined with stereotactic body radiation therapy (SBRT) for patients with oligometastatic esophageal squamous cell carcinoma. Participants will receive anti-PD1 and SBRT to the metastatic lesions which are amenable to the delivery of SBRT after 4~6 cycles of systemic chemotherapy and anti-PD-1.

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group performance status ≤ 2;
2. Histologically confirmed squamous cell carcinoma of the esophagus;
3. Diagnosed with stage IVB disease (according to UICC TNM version 8) with less than five metastatic lesions within three organs;
4. Received 4 to 6 cycles of standard chemotherapy (fluoropyrimidine or taxane-based platinum doublet chemotherapy) and anti-PD1 treatment, and no progression disease was confirmed;
5. At least one metastatic lesions amenable to the delivery of SBRT;
6. Estimated life expectancy >4 months;
7. The function of important organs meet the following requirements: a. white blood cell count (WBC) ≥ 4.0×109/L, absolute neutrophil count (ANC) ≥ 1.5×109/L; b. platelets ≥ 100×109/L; c. hemoglobin ≥ 9g/dL; d. serum albumin ≥ 2.8g/dL; e. total bilirubin ≤ 1.5×ULN, ALT, AST and/or AKP ≤ 2.5×ULN; f. serum creatinine ≤ 1.5×ULN or creatinine clearance rate >60 mL/min;
8. Ability to understand the study and sign informed consent.

Exclusion Criteria:

1. Progression was confirmed after completion of 4 to 6 cycles of standard chemotherapy and anti-PD1 treatment;
2. Patients with intracranial metastasis disease at diagnosis;
3. History of thoracic irradiation;
4. Known or suspected allergy or hypersensitivity to monoclonal antibodies and the chemotherapeutic drugs: Capecitabine, paclitaxel, or platinum;
5. Patients have spinal bone metastases combined with spinal cord compression;
6. A history of malignancies other than esophageal cancer before enrollment, excluding non-melanoma skin cancer, in situ cervical cancer, or cured early prostate cancer;
7. Patients who cannot tolerate radiotherapy due to severe cardiac, lung, liver, or kidney dysfunction, or hematopoietic disease or cachexia;
8. Inability to provide informed consent due to psychological, familial, social, and other factors;
9. Female patients who are pregnant or during lactation;
10. Active autoimmune diseases, a history of autoimmune diseases (including but not limited to these diseases or syndromes, such as colitis, hepatitis, hyperthyroidism), a history of immunodeficiency (including a positive HIV test result), or other acquired or congenital immunodeficiency diseases, a history of organ transplantation or allogeneic bone marrow transplantation;
11. A history of interstitial lung disease or non-infectious pneumonia; Presence of active hepatitis B (HBV DNA ≥ 2000 IU/mL or 104 copies/mL), hepatitis C (positive for hepatitis C antibody, and HCV-RNA levels higher than the lower limit of the assay).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12-10 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
1-year progression-free survival | From date of randomization until the date of death from any cause or the date of first documented disease progression whichever came first, assessed up to 12 months
  1-year progression-free survival

SECONDARY OUTCOMES:
1-year overall survival | From date of randomization until the date of death from any cause or the date of last follow-up, whichever came first, assessed up to 12 months
  1-year overall survival
ORR | 3 months after SBRT (plus or minus 14 days)]
  Overall response rate
Treatment-related adverse events | From the start of treatment to 2 year after the completion of treatment
  Toxicity of treatment was evaluated according to CTCAE 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Mian Xi, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Mian Xi, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu Q, Zhu Z, Chen Y, Deng J, Ai D, Liu Q, Wang S, Wu S, Chen J, Zhao K. Phase 2 Study of Stereotactic Body Radiation Therapy for Patients with Oligometastatic Esophageal Squamous Cell Carcinoma. Int J Radiat Oncol Biol Phys. 2020 Nov 1;108(3):707-715. doi: 10.1016/j.ijrobp.2020.05.003. Epub 2020 May 14. PMID 32417405
- [Background] Liu S, Luo L, Zhao L, Zhu Y, Liu H, Li Q, Cai L, Hu Y, Qiu B, Zhang L, Shen J, Yang Y, Liu M, Xi M. Induction chemotherapy followed by definitive chemoradiotherapy versus chemoradiotherapy alone in esophageal squamous cell carcinoma: a randomized phase II trial. Nat Commun. 2021 Jun 29;12(1):4014. doi: 10.1038/s41467-021-24288-1. PMID 34188053